CLINICAL TRIAL: NCT04888637
Title: Pediatric Language and Memory Mapping in Refractory Epilepsy Using Magnetoencephalography
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 261511
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects: MEG baseline session Receptive Language Task Memory Task
  Interventions: Diagnostic Test: Baseline MEG Test; Behavioral: Receptive Language Task; Behavioral: Memory Task

INTERVENTIONS:
Diagnostic Test: Baseline MEG Test — Each subject will have one MEG session with the recordings of baseline resting state, language and memory protocols. Subjects will have a break period between the language and memory tasks. MEG recordings will be acquired for approximately 35 minutes. The subject will be allowed to practice the language and memory tasks before the MEG recording to feel familiar with them. This practice phase will be a short version of the task administered by a computer and will take approximately 6 minutes.
  Other Names: MEG Acquisition
Behavioral: Receptive Language Task — The subject will perform a practice session where they will be instructed to "try to remember" a set of ﬁve audibly spoken English words, deemed targets (jump, little, please, drink, and good). Depending on the subject's overall verbal memory capacity, the target words will be presented once or twice during the practice phase. Subsequently, during the MEG recording, the ﬁve target words will repeat in a different random order, mixed with a different set of 40 distractors (non-repeating words) in each of three blocks of stimuli. The subject's task will be to listen to the words and lift their index finger of the dominant hand whenever they hear a repeated target word (one of the five). After the language task, the subject will be given a break.
Behavioral: Memory Task — The subject will be tasked with indicating whether the encoding stimulus matched the retrieval stimulus using two buttons; one for "congruent" and the other for "incongruent" response. Button type will be counterbalanced among subjects. The task will take around 16 minutes. The visual stimuli will be projected through an LCD projector onto a white screen located about 0.5 m in front of the subject and subtending 1.0-4.0 and 0.5 degrees of horizontal and vertical visual angle, respectively. A MEG compatible keyboard will be used to measure the subject's responses for "congruent" and "incongruent". The subject will practice the memory task before going to the MEG system using a computer from MEG laboratory. This practice phase will consist of a short version of the memory task with duration of approximately 4 minutes.

SUMMARY:
This is a pilot research study where language and working memory tasks will be used to study brain activities from children with epilepsy. Specifically for language assessment, a well-known MEG language protocol will be used and novel signal processing techniques will be applied. A widely utilized paradigm will be used to study memory function and adapt signal-processing techniques from previous literature for the processing and analysis of MEG signals collected during memory task. No treatment/intervention will be performed or evaluated in this pilot research study.

DETAILED DESCRIPTION:
This is a pilot research study where language and working memory tasks will be used to study brain activities from children with epilepsy. Specifically for language assessment, a well-known MEG language protocol will be used and novel signal processing techniques will be applied. A widely utilized paradigm will be used to study memory function and adapt signal-processing techniques from previous literature for the processing and analysis of MEG signals collected during memory task. No treatment/intervention will be performed or evaluated in this pilot research study.

A MEG scan will be performed and data will be collected from ten pediatric subjects with drug-resistant focal epilepsy under evaluation for resective surgery. If a MRI scan is available from medical records and images have the appropriate characteristics for MEG (see more specifications at MRI section) analysis, MRI will be used for MEG source reconstruction. If MRI is not available, one scan will be performed. MRI is necessary to obtain brain anatomy for high quality MEG source reconstruction.

Quantitative parameters will be extracted from MEG data for evaluating language and memory functions. This is a pilot research study where we will test the feasibility of the recording of both standard language and well-known memory task in patients with epilepsy. This research is important to investigate, by a non-invasive means, possible patterns of language and memory organization that may in future guide surgery and limit potential loss of these functions.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 21 years old
* Drug-resistant focal epilepsy
* Enrolled in the Arkansas Children's Neuroscience Center Comprehensive Epilepsy Program
* Under evaluation for resective surgery
* English speakers. This is not a treatment/intervention study.

Exclusion Criteria:

* Previous resective surgery for epilepsy
* Presence of progressive neurodegenerative disorders
* Presence of significant magnetic artifacts; electronic, magnetic or metallic implants (e.g. pins, screws, shrapnel remains, surgical clips, artificial heart valves, cochlear implants, vascular stents pacemakers); or permanent make-up or tattoos made with metallic dyes
* Presence of seizures within 24 hours of the MEG
* Use of sedation during the MEG acquisition
* Inability to be in a seated or supine position during the tasks
* Major medical disorders (e.g. HIV, cancer)
* Significant visual or auditory disabilities
* Physical disabilities that interfere with accomplishment of study tasks (when applicable)
* Claustrophobia, or fear of cramped or confined spaces
* Pregnancy or suspected pregnancy
* Any condition that the investigator feels might put the patient at risk

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of fifteen (15) pediatric patients with drug-resistant focal epilepsy under evaluation for resective surgery will be recruited from the comprehensive epilepsy program of the Arkansas Children's Neuroscience Center. If the patient is eligible, they will be informed about this study during their routine clinic visits by their clinician, and asked if they are interested in participating. Those who express an interest will be provided with the informed consent form (ICF) approved by the UAMS Institutional Review Board (IRB).
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana I Escalona-Vargas, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 pediatric patients with drug-resistant focal epilepsy were recruited from the comprehensive epilepsy program of the Arkansas Children's Neuroscience Center
Pre-assignment Details: Only one group: epilepsy group
Groups:
- All Subjects: only one group: epilepsy group
Period: Overall Study
Arm/Group | All Subjects
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 8-21 years of age
Groups:
- All Subjects. This is Not a Treatment/Intervention Study.: This is not a treatment/intervention study. Thus, we don't have comparison groups. Participants were not assigned into Participant Flow or intervention strategy.
Arm/Group | All Subjects. This is Not a Treatment/Intervention Study.
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Completed MEG
Description: This is not a treatment/intervention study. Pilot study was to record brain activity utilizing a noninvasive MEG system during resting state, receptive language and working memory tasks.
Time Frame: only one measurement in one visit
Population: We were able to record brain activity utilizing a noninvasive MEG system during resting state, receptive language and working memory tasks in 10 children with epilepsy. 1 MEG per subject enrolled
Measure: Number; unit: participants
Groups:
- All Subjects: epilepsy
Arm/Group | All Subjects
Number analyzed (Participants) | 10
participants | 1

ADVERSE EVENTS:
Time Frame: 30 days
Description: The definition of Adverse event and/or serious adverse event does not differ from the clinicaltrials.gov definition.
Groups:
- All Subjects: only one group: epilepsy
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04888637/Prot_SAP_000.pdf